CLINICAL TRIAL: NCT05580367
Title: Gut-Brain-Axis/Lung-Brain-Axis and Mental Ill Health in Critical Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0428
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Mental Health Issue; Critical Illness; Gut Microbiome
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survivors of critical illness commonly experience long-lasting cognitive, mental health and physical impairments. Clinically significant symptoms of anxiety, depression, and post-traumatic stress disorder (PTSD) may occur in 40%, 34% and 20% of ICU survivors respectively, compared to 6%, 8% and 4% in the general population. These symptoms can persist for more than 8 years.

Evidence shows the existence of a two-way, communication network between gut microbes and the brain referred to as the gut-brain axis. Changes in the microbiome and dysregulation of this communication network in relatively healthy people is associated with cognitive dysfunction and mood disorders such as anxiety and depression. The physiological stress associated with critical illness itself and many ICU interventions including the use of mechanical ventilation and medications such as antibiotics, antacids, vasopressors, and steroids can influence the balance of the gut microbiome and associated metabolites.

This observation study aims to:

1. Quantify and measure dynamic changes in the gut microbiome and its metabolites during critical illness and recovery.
2. Explore the associations between microbiome and metabolomic changes during critical illness and psychological symptoms in the patient during their recovery.

This knowledge will provide the potential to create interventions that alter the gut environment and microbiome both during and following a critical illness in order to reduce long-term adverse psychological effects. Examples of such potential interventions include dietary modifications with the use of prebiotics or probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Unplanned admission to critical care
* Aged ≥18 years old
* Requiring mechanical ventilation
* Commencing ventilation within the previous 24 hours
* Expected to be ventilated for minimum of ≥72 hours

Exclusion Criteria:

* Known prior diagnosis of cognitive impairment
* Known prior mental ill health
* Known malignancy
* Admitted after presenting with any of the following conditions:
* trauma
* brain injury
* surgery
* cardiac arrest
* immunosuppressed
* underlying pyogenic infection
* Not expected to survive to completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an unplanned admission to critical care who are mechanically ventilated
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome changes | 3 months post-discharge
  Quantify and measure dynamic changes in the gut microbiome and its metabolites during critical illness and recovery. (The number and diversity of microbe present)
Microbiome, metabolic changes and psychological symptoms | 3 months post-discharge
  Explore the associations between microbiome and metabolomic changes during critical illness and psychological symptoms in the patient during their recovery.
Gut microbial and metabolic signatures | 3 months post-discharge
  Investigate the potential for gut microbial and metabolic signatures at admission and discharge to predict the future development of psychological symptoms following ICU discharge.
Sample repository | 3 months post-discharge
  Establish a sample repository for future analysis for future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom